CLINICAL TRIAL: NCT03396003
Title: GALILEI G6 Lens Professional vs. a Predicate Device: a Comparison Study
Brief Title: A Comparison of Two Devices for Taking Measurements of the Eye to Assist in Lens Selection for Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZIEMER_G6
Record Dates: First submitted 2017-11-20; First posted 2018-01-10 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- GALILEI G6 Lens Professional (Experimental): The GALILEI G6 Lens Professional will measure anterior segment geometry and axial intra-ocular distances of the eye.
  Interventions: Device: GALILEI G6 Lens Professional
- Oculus Pentacam AXL (Active Comparator): The Oculus Pentacam AXL will measure anterior segment geometry and axial intra-ocular distances of the eye.
  Interventions: Device: Oculus Pentacam AXL

INTERVENTIONS:
Device: GALILEI G6 Lens Professional — Eight measurements of the eye using the GALILEI G6 Lens Professional will be taken using two different devices and 2 different operators
  Arms: GALILEI G6 Lens Professional
Device: Oculus Pentacam AXL — A single measurement of the eye will be taken using the Oculus Pentacam AXL
  Arms: Oculus Pentacam AXL

SUMMARY:
The purpose of this study is to compare the Ziemer Ophthalmic Systems AG GALILEI G6 Lens Professional to the Oculus Pentacam® AXL for taking images and measurements of the anterior segment of the eye, including the cornea, pupil, anterior chamber and lens, to assist in determining the power of the intraocular lens for implantation.

DETAILED DESCRIPTION:
A corneal topographer/biometer named GALILEI G6 Lens Professional was developed by Ziemer Ophthalmic Systems AG for the measurement of anterior segment geometry and axial intraocular distances. The measurement principle of the corneal topographer corresponds to that of the commercially available Galilei G4 Dual Scheimpflug Analyzer, whereas the measurement principle of the biometer is based on low coherence interferometry/reflectometry, which has been widely used and applied clinically by a number of predicate devices.

One complete measurement consists of a corneal topography/ tomography scan followed by three consecutive, axial biometry scans of the anterior segment (cornea and crystalline lens) and three consecutive, axial biometry scans of the retina. The measurement process is continuous but divided into three alignment-click-steps.

Such measurements can be applied to given Intra Ocular Lens (IOL) types and IOL equations, to permit the calculation of recommended IOLs to be implanted during cataract surgery in order to achieve the desired vision correction.

The primary objectives of this clinical study are to: 1) evaluate the inter-device repeatability, inter-operator repeatability and reproducibility of the GALILEI G6 Lens Professional in repeated measurements of anterior segment geometry and axial intraocular distances and, 2) demonstrate substantial equivalence through examining agreement of the GALILEI measurements to those of the predicate device, the Pentacam® AXL.

ELIGIBILITY:
Inclusion Criteria:

* Satisfies one of the subject group categories and the enrollment quota for that category has not been reached:

  1. Normal eyes (phakic eyes without cataracts or corneal disease, refraction ≥ -5.5 D or ≤ +5.0 D)
  2. Eyes having undergone previous refractive surgery (LASIK or PRK)
  3. Eyes with cataracts (LOCS III grading with grades 2-6 in any or all of the posterior subcapsular (P2-P5), nuclear (N2-N5) and cortical (C2-C5), assessed by slit lamp examination; no other known ocular pathology)
  4. Eyes with severe myopia (≤ -6 D according to the American Academy of Ophthalmology)
  5. Eyes with severe hyperopia (≥ +5.25 D according to the American Academy of Ophthalmology)
  6. Eyes with previous cross-linking and eyes with advanced keratoconus
* Manifest refraction sSpherical eEquivalent Refraction (MRSER) between -10dpt and +10dpt as measured by cycloplegic autorefraction assessed less than 12 months prior to enrollment
* Best corrected visual acuity (BCVA) of LogMAR 0.2 or better

Exclusion Criteria:

* Strabismus, nystagmus, amblyopia, anisometropia (difference in MRSER>3D)
* Angle closure glaucoma
* Seizure disorder, brain damage, Down Syndrome, Trisomy 13 or 18, Cerebral Palsy or other serious ophthalmic or central nervous system disorders
* Severe dry eye
* Severe corneal scarring
* Inability to hold gaze
* Inability to see fixation target

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Axial Length (AL) Measurement in millimeters (mm) | One day
  Repeatability and reproducability across and between evaluations
Central Corneal Thickness (CCT) Measurement in micrometers (µm) | One day
  Repeatability and reproducability across and between evaluations
Radius Flat Meridian (R flat) Measurement in millimeters (mm) | One day
  Repeatability and reproducability across and between evaluations
Radius Steep Meridian (R steep) Measurement in millimeters (mm) | One day
  Repeatability and reproducability across and between evaluations
Mean Radius (Rm) Measurement in millimeters (mm) | One day
  Repeatability and reproducability across and between evaluations
Corneal Cylinder Measurement in diopters (D) | One day
  Repeatability and reproducability across and between evaluations
Corneal Cylinder Axis (A flat) Measurement in degrees | One day
  Repeatability and reproducability across and between evaluations
Anterior Chamber Depth (ACD) Measurement in millimeters (mm) | One day
  Repeatability and reproducability across and between evaluations
Horizontal White-to-White distance (WtW) Measurement in millimeters (mm). | One day
  Repeatability and reproducability across and between evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Majid Moshirfar, MD, Principal Investigator
Locations (1):
- Ziemer Ophthalmic Systems AG, Port, Switzerland

IPD SHARING:
Plan to Share IPD: No